CLINICAL TRIAL: NCT00383773
Title: Retinal Endo Vascular Surgery for Central Retinal Vein Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1yumbo-HMO-CTIL
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-09

CONDITIONS: Central Retinal Vein Occlusion
Keywords: retinal vein occlusion; rTPA
MeSH Terms: conditions — Retinal Vein Occlusion

INTERVENTIONS:
Procedure: Retinal endo vascular surgery

SUMMARY:
Patients with Central Retinal Vein Occlusion will undergo vitrectomy, a small needle of about 71 micron will enter a branch retinal vein and TPA will be injected into the obstracted vein.

DETAILED DESCRIPTION:
Patients with Central Retinal Vein Occlusion less than 6 month duration and reduction of vision to 6/21 will go OCT and FANG examinations.

Patient will be operated vitrectomy, and a branch retinal vein will be punctured by small needle and rTPA 200mcg/ml will be injected to the vein.

ELIGIBILITY:
Inclusion Criteria:

* crvo less than 6 month
* Visual Acuity less than 6/21
* No prior eye surgery except cataract.

Exclusion Criteria:

* Retinal/iris neovascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-10; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Visual acuity
Amount of macular edema.

CONTACTS AND LOCATIONS:
Overall Officials: Michael halpert, Study Chair — Hadassah Medical Organization